CLINICAL TRIAL: NCT03677518
Title: Total Knee Arthroplasty With the Medial-Pivot Knee System: Clinicaland Radiological Outcomes at 9.5 Years' Mean Follow-up
Brief Title: Total Knee Arthroplasty With the Medial-Pivot Knee System
Acronym: MEDIAL-PIVOT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0052
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-09

CONDITIONS: Arthroplasty Complications
Keywords: total knee arthroplasty; medial-pivot knee system; kinematics; survivorship

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The "ball-in-socket" design of the Medial-Pivot knee system (MicroPort Orthopedics, Arling-ton, Tennessee, USA) aims to reproduce normal knee kinematics by medializing its rotational axis. Thegoal of this study was to measure knee range of motion (ROM) with this implant after a mean follow-up of 10 years and to report the survivorship and long-term clinical and radiological outcomes. Wehypothesized the prosthetic knee would have at least 120◦flexion at 10 years. This was retrospective, single-centre study of 74 Medial-Pivot knees implanted in71 patients (average age of 69 years) between May 2005 and November 2007. All patients who receiveda Medial-Pivot knee were included consecutively. The mean follow-up was 10 years. Clinical and radio-logical assessments were performed using the Knee Society Score (KSS) and Ewald's score. Kaplan-Meirsurvival analysis was used to calculate survivorship.

DETAILED DESCRIPTION:
methodsThis was retrospective, single-centre study of 74 Medial-Pivotknees implanted in 71 patients between May 2005 and Novem-ber 2007. During this period, several types of semi-constrainedprimary TKA implants were used.The "ball-in-socket" design of the Medial-Pivot knee system (MicroPort Orthopedics, Arling-ton, Tennessee, USA) aims to reproduce normal knee kinematics by medializing its rotational axis. Thegoal of this study was to measure knee range of motion (ROM) with this implant after a mean follow-up of 10 years and to report the survivorship and long-term clinical and radiological outcomes. Wehypothesized the prosthetic knee would have at least 120◦flexion at 10 years. This was retrospective, single-centre study of 74 Medial-Pivot knees implanted in71 patients (average age of 69 years) between May 2005 and November 2007. All patients who receiveda Medial-Pivot knee were included consecutively. The mean follow-up was 10 years. Clinical and radio-logical assessments were performed using the Knee Society Score (KSS) and Ewald's score. Kaplan-Meirsurvival analysis was used to calculate survivorship.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years
* patienst must be operated
* patient with mid-line skin incision

Exclusion Criteria:

* patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were operated by four experienced surgeons usingthe same protocol. A mid-line skin incision was made in all patientsexcept one who had previously undergone a lateral osteotomy. The parapatellar arthrotomy was medial in all cases. Independent tibialand femoral cuts were made with an intramedullary femoral aim-ing device targeting 7◦valgus in 48 cases and 5◦in 2 cases. Femoral component external rotation of 3◦relative to the posterior condy-lar plane was applied in all patients. All implants were fixed usingPalacos®bone cement with gentamicin (Haeraus, Warsaw, USA).The patella was resurfaced in 40 knees.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Flexion with an Advance® Medial-Pivot knee | 2years
  The objective of this study was to evaluate the flexion in patients with an Advance® Medial-Pivot knee after an average follow-upof 10 years. Knee flexion was measured with a goniometer in the office; thegreater trochanter, knee centre and lateral malleolus were used asreference points.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Mertl, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No